CLINICAL TRIAL: NCT03599674
Title: Targeted Inpatient Navigation to Improve Care for Minority Children and Families
Acronym: TNav
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Responsible Party: Principal Investigator, K. Casey Lion, Investigator | Center for Child Health, Behavior and Development, Seattle Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00000852
Record Dates: First submitted 2018-06-04; First posted 2018-07-26 (Actual); Last update posted 2021-06-25 (Actual); Status verified 2021-06

CONDITIONS: Hospitalized Children

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Family Bridge Program (Experimental): Families receive Family Bridge Program services which include orientation to the hospital, concrete needs assessment, communication preferences assessment, communication coaching, follow-up during the hospital stay, and a follow-up phone call after discharge.
  Interventions: Behavioral: Family Bridge Program

INTERVENTIONS:
Behavioral: Family Bridge Program — Families receive Family Bridge Program services which include orientation to the hospital, concrete needs assessment, communication preferences assessment, communication coaching, follow-up during the hospital stay, and a follow-up phone call after discharge.

SUMMARY:
The overall goal of this research is to evaluate a new program designed to address basic human needs, create a safe and supportive environment for families, and help families build skills and confidence for navigating the health care system.

Specifically, we aim to pilot test the feasibility and acceptability of the Targeted Inpatient Navigation (TNav) program for families of low income, minority hospitalized children.

ELIGIBILITY:
Inclusion Criteria:

* Caregiver ≥18 years of age, with a hospitalized child <18 years old
* Preferred language of English, Spanish and Somali
* child with Medicaid insurance or no insurance
* child with self-reported (or parent-reported) minority race/ethnicity
* within 3 days of admission/ transfer to the medical unit on a general medicine service of a resident team

Exclusion Criteria:

* Admission for suspected child abuse
* Involvement of Child Protective Services at time of admission
* Admission for primary mental health condition, including intentional ingestion and eating disorder
* Family already enrolled in longer-term navigation services

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-04-16 (Actual); Primary Completion 2018-10-19 (Actual); Study Completion 2018-10-29 (Actual)

PRIMARY OUTCOMES:
Program acceptability to caregivers--qualitative | 4-6 weeks after discharge
  Program acceptability will be determined qualitatively, on the basis of thematic content analysis of semi-structured interviews with enrolled caregivers
Program feasibility | Calculated for each family after program involvement is complete, generally 1 week after discharge.
  Ability to deliver program elements as planned, calculated as the number of Family Bridge services delivered to a family divided by the services available to that family.
Program acceptability to providers--qualitative | Once per month, every month that they care for an enrolled family, up to 6 months
  Program acceptability will be determined qualitatively, on the basis of thematic content analysis of semi-structured interviews with the doctors, nurses, social workers and care coordinators who were involved in their hospital care.

SECONDARY OUTCOMES:
Cultural Distance Scale | Enrollment and 2-4 weeks after discharge.
  4 items measuring perceived similarity or difference in norms and values between family and medical providers. Each of the 4 items is scored on a Likert scale from 1 to 6, with higher values reflecting greater difference. The total scale score is the average of the 4 responses, on a scale from 1 to 6.
Barriers to Care Questionnaire | Enrollment and 2-4 weeks after discharge.
  20 items measuring perceived barriers to medical care, with 4 sub-scales, each scored and reported separately: System as a whole, Skills barriers, Expectation barriers, and Knowledge barriers. Each subscale was scored 0-100, with higher scores indicating greater barriers.
Perceived Efficacy in Patient-Physician Interactions (PEPPI) | Enrollment and 2-4 weeks after discharge.
  10-item tool measuring understanding of and ability to interact with health professionals and organizations.
Perceived Stress Scale-short form | Enrollment and 2-4 weeks after discharge.
  4 items, scored from 0 (Never) to 4 (Very Often), related to perceived stress and control over one's life. Responses are summed for a total score from 0 to 16, with higher scores reflecting greater stress.
Local system navigation | Enrollment and 2-4 weeks after discharge.
  9 items assessing familiarity with navigating the local health care system.
Communication--Pediatric H-CAHPS | 2-4 weeks after discharge.
  9 items assessing quality of communication from doctors and nurses, including at discharge.
Partnership--Pediatric H-CAHPS | 2-4 weeks after discharge.
  3 items assessing provider-family partnership.
Health care transition questions | 2-4 weeks after discharge.
  10 items assessing quality of transition and comfort and understanding of home care.
Unmet need for navigation | 2-4 weeks after discharge.
  7 items to determine whether family's needs were identified and met during hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: K.Casey Lion, MD, MPH, Principal Investigator — Seattle Children's Hospital
Locations (1):
- Seattle Children's Hospital, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lion KC, Arthur KC, Frias Garcia M, Hsu C, Sotelo Guerra LJ, Chisholm H, Griego E, Ebel BE, Penfold RB, Rafton S, Zhou C, Mangione-Smith R. Pilot Evaluation of the Family Bridge Program: A Communication- and Culture-Focused Inpatient Patient Navigation Program. Acad Pediatr. 2024 Jan-Feb;24(1):33-42. doi: 10.1016/j.acap.2023.06.021. Epub 2023 Jun 22. PMID 37354947
- [Derived] Chisholm H, Kershaw T, Sotelo Guerra L, Bocek K, Garcia Y, Lion KC. A Realist Evaluation Analysis of a Novel Multi-Faceted Inpatient Patient Navigation Program. Acad Pediatr. 2022 Jul;22(5):789-796. doi: 10.1016/j.acap.2021.09.009. Epub 2021 Sep 20. PMID 34551342